CLINICAL TRIAL: NCT00969761
Title: A Phase I Dose Escalation Trial of BI 6727 in Combination With Cisplatin or Carboplatin in Patients With Advanced or Metastatic Solid Tumors
Brief Title: BI 6727 (Volasertib) in Combination With Cisplatin or Carboplatin in Patients With Advanced or Metastatic Solid Tumour
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1230.6; 2008-003926-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727

ARMS (2):
- A. BI 6727-cisplatin (Experimental): patient to receive 3-weekly infusion escalating dose of BI 6727 combined to cisplatin
  Interventions: Drug: BI 6727
- B. BI 6727-carboplatin (Experimental): patient to receive 3-weekly infusion escalating dose of BI 6727 combined to carboplatin
  Interventions: Drug: BI-6727

INTERVENTIONS:
Drug: BI-6727 — Low to high dose (administered every 3 weeks). Depending on the toxicities observed, intermediary dose levels may be added
  Arms: B. BI 6727-carboplatin
Drug: BI 6727 — low to high dose
  Arms: A. BI 6727-cisplatin

SUMMARY:
The primary objective of this trial is to identify the maximum tolerated dose (MTD) of BI 6727 therapy in terms of drug-related adverse events when combined with a platinum therapy (cisplatin or carboplatin).

Secondary objectives are the collection of overall safety and antitumour efficacy data and the determination of the pharmacokinetic profile of BI 6727 combination treatment with cisplatin and carboplatin.

ELIGIBILITY:
Inclusion criteria:

1. Patients with confirmed diagnosis of advanced, non resectable and / or metastatic solid tumours, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment
2. Indication for a treatment with platinum therapy as judged by the investigator
3. Age 18 years or older
4. Written informed consent consistent with ICH-GCP and local legislation
5. ECOG performance score lower or equal 2
6. Recovery from CTCAE Grade 2 - 4 therapy-related toxicities from previous systemic anti-cancer therapies or radiotherapies (except alopecia grade 2)

Exclusion criteria:

1. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
2. Pregnancy or breastfeeding
3. Active infectious disease or known chronic Hepatitis B/Hepatitis C infection and HIV I/II
4. Clinical evidence of symptomatic progressive brain or leptomeningeal disease during the past 6 months
5. Second malignancy currently requiring another anti-cancer therapy
6. ANC less than 1500 / mm3
7. Platelet count less than 100 000 / mm3
8. Bilirubin greater than 1.5 mg / dl (> 26 micromol / L, SI unit equivalent) (except Gilbert's syndrome)
9. Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
10. Serum creatinine greater than 1.5 mg / dl (> 132 micromol / L, SI unit equivalent) or creatinine clearance <70ml/min (as calculated according to Cockcroft-Gault formula for GFR estimate)
11. Known history of relevant QT-prolongation, e.g. long QT-syndrome
12. Pre-existing clinically relevant hearing loss
13. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
14. Treatment with other investigational drugs or participation in another clinical interventional trial within the past four weeks before start of therapy or concomitantly with this trial
15. Systemic anti-cancer therapy or radiotherapy within the past four weeks before start of therapy or concomitantly with this trial. This restriction does not apply to steroids and bisphosphonates.
16. Patients unable to comply with the protocol
17. Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Belgium (2):
  - 1230.6.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1230.6.3202 Boehringer Ingelheim Investigational Site, Leuven

REFERENCES:
- [Derived] Awada A, Dumez H, Aftimos PG, Costermans J, Bartholomeus S, Forceville K, Berghmans T, Meeus MA, Cescutti J, Munzert G, Pilz K, Liu D, Schoffski P. Phase I trial of volasertib, a Polo-like kinase inhibitor, plus platinum agents in solid tumors: safety, pharmacokinetics and activity. Invest New Drugs. 2015 Jun;33(3):611-20. doi: 10.1007/s10637-015-0223-9. Epub 2015 Mar 22. PMID 25794535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, parallel group, 3+3 dose escalation trial Volasertib and cisplatin or carboplatin combination therapy was given on Day 1 of up to 6, 3-week cycles.
Pre-assignment Details: For the carboplatin arm, the target doses were calculated using the Calvert formula to achieve AUC 4, AUC 5 and AUC 6. Calvert formula: Dose (mg) = target AUC x (glomerular filtration rate (GFR) + 25); GFR = (140 - age [years]) x (actual weight [kg])/(72 x serum creatinine [mg/dL]). Multiply by another factor of 0.85 if female).
Groups:
- V200+Cis75: Patients received 200mg Volasertib (V200) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus 75mg/m2 cisplatin (Cis) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V300+Cis75: Patients received 300mg Volasertib (V300) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus 75mg/m2 cisplatin (Cis) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V300+Cis100: Patients received 300mg Volasertib (V300) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus 100mg/m2 cisplatin (Cis) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V350+Cis75: Patients received 350mg Volasertib (V350) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus 75mg/m2 cisplatin (Cis) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V100+Car4: Patients received 100mg Volasertib (V100) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus AUC4 (area under the curve of 4) carboplatin (Car) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V100+Car5: Patients received 100mg Volasertib (V100) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus AUC5 (area under the curve of 5) carboplatin (Car) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V200+Car5: Patients received 200mg Volasertib (V200) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus AUC5 (area under the curve of 5) carboplatin (Car) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V300+Car5: Patients received 300mg Volasertib (V300) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus AUC5 (area under the curve of 5) carboplatin (Car) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V300+Car6: Patients received 300mg Volasertib (V300) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus AUC6 (area under the curve of 6) carboplatin (Car) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V350+Car5: Patients received 350mg Volasertib (V350) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus AUC5 (area under the curve of 5) carboplatin (Car) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V100+Cis60: Patients received 100mg Volasertib (V100) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus 60mg/m2 cisplatin (Cis) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
- V100+Cis75: Patients received 100mg Volasertib (V100) administered by intravenous infusion over 2 hours at day 1 of each treatment cycle, plus 75mg/m2 cisplatin (Cis) administered by intravenous infusion over 1 hour at day 1 of each treatment cycle.
Period: Discont. Before Start of Treat. Cycle 2
Arm/Group | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5 | V100+Cis60 | V100+Cis75
Started | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3 | 3 | 3
Completed | 2 | 3 | 10 | 5 | 3 | 3 | 3 | 6 | 11 | 2 | 3 | 3
Not Completed | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Dose Limiting Toxicity (DLT) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other adverse events | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Treated in and Beyond Treat. Cycle 2
Arm/Group | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5 | V100+Cis60 | V100+Cis75
Started | 2 | 3 | 10 | 5 | 3 | 3 | 3 | 6 | 11 | 2 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 10 | 5 | 3 | 3 | 3 | 6 | 11 | 2 | 3 | 3
Not completed — Progressive disease | 2 | 3 | 10 | 3 | 2 | 3 | 3 | 6 | 9 | 2 | 3 | 3
Not completed — Other adverse events | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients who received at least one administration of volasertib and cisplatin or carboplatin.
Groups:
- Total: Total of all reporting groups
Arm/Group | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5 | V100+Cis60 | V100+Cis75 | Total
Number analyzed (Participants) | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3 | 3 | 3 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (7.51) | 55.0 (12.53) | 52.5 (16.67) | 60.0 (9.53) | 56.3 (11.72) | 54.0 (5.57) | 58.0 (13.75) | 66.3 (10.07) | 51.8 (13.03) | 58.3 (6.66) | 45.0 (19.16) | 58.3 (7.37) | 54.7 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 2 | 1 | 1 | 1 | 2 | 6 | 2 | 2 | 2 | 27
  Male | 0 | 1 | 9 | 4 | 2 | 2 | 2 | 4 | 7 | 1 | 1 | 1 | 34

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The maximum tolerated dose (MTD) was defined as the highest dose studied for which the incidence of DLT was less than 33% (i.e. 1/6 patients) during the first cycle, for Volasertib in combination with cisplatin or carboplatin.
  0=not maximum tolerated dose, 1=was maximum tolerated dose.
Time Frame: 3 weeks
Population: Treated set
Measure: Number; unit: Units on a scale
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Units on a scale | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: Percentage of Participants With Dose Limiting Toxicities
Description: Percentage of participants with dose limiting toxicities (DLTs) during the first treatment cycle.
Time Frame: 3 weeks
Population: Treated set.
  There was one patient in the V300+Car6 group whose DLT data was not evaluable, so only 12 patients had evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 25.0 | 33.3 | 0.0 | 0.0 | 0.0 | 16.7 | 16.7 | 66.7

3. Secondary Outcome: Objective Response Rate
Description: Objective response was defined as the proportion of participants having at least a best response of complete response (CR) or partial response (PR) determined based on RECIST criteria, version 1.0 (V1.0).
  Tumour response was documented using appropriate techniques
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants | 0.0 | 33.3 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 7.7 | 0.0

4. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response was defined as the time from first documented confirmed complete response (CR) or partial response (PR) to first evidence of progressive disease (PD) or death from any cause, whichever occurred first, determined based on RECIST V1.0 criteria.
  Tumour response was documented using appropriate techniques
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set restricted to participants with confirmed objective response.
Measure: Median (Full Range); unit: Days
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Days |  | 298 [298 to 298] |  | 359 [359 to 359] |  |  |  |  |  | 282 [282 to 282] | 207 [207 to 207] |

5. Secondary Outcome: Best Overall Response
Description: Best overall response was defined as the best response obtained since the start of study treatment until disease progression, determined based on RECIST V1.0 criteria.
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants
  Complete response | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Partial response | 0.0 | 33.3 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 7.7 | 0.0
  Stable disease | 66.7 | 66.7 | 33.3 | 33.3 | 25.0 | 33.3 | 33.3 | 33.3 | 0.0 | 33.3 | 7.7 | 33.3
  Progressive disease | 33.3 | 0.0 | 33.3 | 33.3 | 58.3 | 50.0 | 66.7 | 66.7 | 100.0 | 33.3 | 61.5 | 33.3
  Non evaluable | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0
  No post-baseline tumour assessment | 0.0 | 0.0 | 33.3 | 0.0 | 16.7 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 23.1 | 33.3

6. Secondary Outcome: Disease Control Rate
Description: Percentage of participants with confirmed disease control, defined as the proportion of patients with a best overall response of at least stable disease (SD), determined based on RECIST V1.0 criteria.
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants | 66.7 | 100.0 | 33.3 | 66.7 | 25.0 | 33.3 | 33.3 | 33.3 | 0.0 | 50.0 | 15.4 | 33.3

7. Secondary Outcome: Duration of Disease Control
Description: Duration of Disease control was defined as the time from the start of study treatment to the time of disease progression or death, whichever occurred first.
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set restricted to participants with confirmed disease control.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 2 | 3 | 1 | 2 | 3 | 2 | 1 | 1 | 0 | 3 | 2 | 1
Days | 196.5 (103.94) | 309.0 (105.93) | 264.0 (NA) — Not calculable as data only available for one patient | 268.0 (237.59) | 155.0 (49.36) | 103.5 (9.19) | 135.0 (NA) — Not calculable as data only available for one patient | 229.0 (NA) — Not calculable as data only available for one patient |  | 234.0 (115.99) | 190.5 (74.25) | 126.0 (NA) — Not calculable as data only available for one patient

8. Secondary Outcome: Progression-free Survival
Description: Progression-free survival based on RECIST V1.0 criteria was defined as the time from start of treatment to the date of evidence of progressive disease (PD) or death from any cause, whichever occurred first.
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Median (Full Range); unit: Days
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Days | 123.0 [38 to 270] | 309.0 [143 to 340] | 37.0 [1 to 264] | 100.0 [43 to 436] | 49.5 [1 to 232] | 69.5 [21 to 169] | 80.0 [37 to 135] | 64.0 [36 to 229] | 40.0 [36 to 43] | 71.0 [38 to 331] | 43.0 [1 to 243] | 39.0 [13 to 126]

9. Secondary Outcome: Incidence and Intensity of Adverse Events According to CTCAE Version 3.0
Description: Incidence and intensity of adverse events according to common terminology criteria for adverse events (CTCAE) version 3.0
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants
  Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Grade 2 | 0.0 | 0.0 | 66.7 | 33.3 | 8.3 | 16.7 | 0.0 | 33.3 | 66.7 | 0.0 | 0.0 | 0.0
  Grade 3 | 100.0 | 100.0 | 33.3 | 0.0 | 41.7 | 50.0 | 66.7 | 66.7 | 33.3 | 50.0 | 61.5 | 33.3
  Grade 4 | 0.0 | 0.0 | 0.0 | 66.7 | 41.7 | 33.3 | 0.0 | 0.0 | 0.0 | 50.0 | 23.1 | 66.7
  Grade 5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 15.4 | 0.0

10. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: Percentage of participants with serious adverse events (AEs)
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants | 66.7 | 33.3 | 0.0 | 33.3 | 50.0 | 50.0 | 33.3 | 0.0 | 33.3 | 16.7 | 46.2 | 66.7

11. Secondary Outcome: Percentage of Participants With Significant Adverse Events
Description: Percentage of participants with significant adverse events (AEs): dose limiting toxicity (DLT) was defined as significant AE.
  DLTs (i.e. significant AEs) per protocol were:
  * drug related CTCAE grade 3 or 4 non haematological toxicity (except vomiting or diarrhoea responding to supportive treatment and ototoxicity)
  * drug related CTCAE grade 4 neutropenia for seven or more days and / or complicated by infection
  * drug related CTCAE Grade 4 thrombocytopenia
  * drug related febrile neutropenia grade 3 (ANC<1000/mm³ and fever≥ 38.5°C)
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants | 0.0 | 0.0 | 0.0 | 66.7 | 25.0 | 33.3 | 0.0 | 0.0 | 0.0 | 16.7 | 15.4 | 0.0

12. Secondary Outcome: Total Plasma Clearance After Intravascular Administration (CL)
Description: Total plasma clearance after intravascular administration (CL) of Volasertib in combination with cisplatin or carboplatin during treatment cycle 1.
Time Frame: 1 hour (h) 35 minutes (min) before start of volasertib infusion and 1h, 2h, 8h, 24h, 48h, 168h and 336h after start of volasertib infusion
Population: Pharmacokinetic (PK) set which included all participants in the treated set with evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 11 | 6 | 3 | 3 | 3 | 6 | 10 | 3
mL/min | 852 (28.1) | 1130 (28.1) | 1090 (7.60) | 1050 (22.7) | 971 (28.6) | 1010 (47.9) | 1110 (33.6) | 812 (11.7) | 881 (6.92) | 808 (20.7) | 974 (19.1) | 546 (16.7)

13. Secondary Outcome: Apparent Volume of Distribution at Steady State Following Intravascular Administration (Vss)
Description: Apparent volume of distribution at steady state following intravascular administration (Vss) of Volasertib in combination with cisplatin or carboplatin during treatment cycle 1.
Time Frame: as for outcome 12
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 11 | 6 | 3 | 3 | 3 | 6 | 10 | 3
Litres | 6580 (66.9) | 11100 (20.1) | 5570 (18.9) | 7140 (42.5) | 5880 (67.6) | 7270 (41.5) | 8810 (38.7) | 9960 (44.7) | 8950 (36.9) | 8270 (42.2) | 7440 (31.9) | 3640 (35.9)

14. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from baseline in pulse rate at last value on treatment
Time Frame: Baseline and from first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
bpm | 10.0 (10.00) | 23.3 (15.01) | 6.7 (17.24) | -11.7 (14.29) | 10.3 (14.35) | 5.2 (10.34) | 3.7 (26.50) | 0.7 (7.37) | 12.0 (7.55) | 5.7 (10.61) | 14.4 (10.97) | -21.7 (17.79)

15. Secondary Outcome: Change From Baseline in Neutrophils
Description: Change from baseline in neutrophils with the maximum value on treatment
Time Frame: Baseline and from first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Mean (Standard Deviation); unit: 10^9 cells /L
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
10^9 cells /L | 7.6 (7.3) | 3.3 (1.9) | 3.4 (2.3) | 3.0 (2.6) | 6.0 (4.3) | 5.2 (6.5) | 2.1 (3.1) | 6.8 (8.2) | 3.6 (2.7) | 5.9 (6.9) | 5.5 (2.4) | 4.7 (2.8)

16. Secondary Outcome: Change From Baseline in Platelets
Description: Change from baseline in platelets with the maximum value on treatment
Time Frame: Baseline and from first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Mean (Standard Deviation); unit: 10^9 cells /L
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
10^9 cells /L | 57 (48) | 65 (78) | 96 (94) | 71 (58) | 67 (58) | 89 (95) | 186 (96) | 50 (38) | 49 (65) | 39 (20) | 73 (58) | 104 (53)

17. Secondary Outcome: Frequency of Participants (%) With Possible Clinically Significant Abnormalities for Neutrophils
Description: Frequency of participants (%) with possible clinically significant abnormalities for neutrophils: : defined as neutrophils >=CTCAE grade 2 (CTCAE v3.0), with worsening from baseline. The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE).
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants | 33.0 | 100.0 | 0.0 | 66.7 | 75.0 | 50.0 | 33.3 | 33.3 | 33.3 | 83.3 | 76.9 | 100.0

18. Secondary Outcome: Frequency of Participants (%) With Possible Clinically Significant Abnormalities for Platelets
Description: Frequency of participants (%) with possible clinically significant abnormalities for platelets : defined as platelets >=CTCAE grade 2 (based on CTCAE v3.0), with worsening from baseline.
  The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE).
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants | 0.0 | 0.0 | 0.0 | 33.0 | 41.7 | 83.3 | 0.0 | 33.3 | 0.0 | 83.3 | 76.9 | 100.0

19. Secondary Outcome: Frequency of Participants With Transitions Relative to the Baseline CTC Grade for Platelets Based on Last Value on Treatment
Description: Percentage of participants with transitions relative to the baseline CTC grade (version 3) for platelets based on last value on treatment.
  Common terminology criteria for adverse events (CTCAE) grade on treatment for platelets (CTC version 3). The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE).
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants
  Baseline=0, last value=0 | 33.3 | 66.7 | 100.0 | 100.0 | 83.3 | 100.0 | 100.0 | 66.7 | 66.7 | 83.3 | 84.6 | 100.0
  Baseline=0, last value=1 | 33.3 | 33.3 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0 | 33.3 | 33.3 | 0.0 | 7.7 | 0.0
  Baseline=1, last value=0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Baseline=0, last value=2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 7.7 | 0.0
  Baseline=0, last value=3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Baseline=1, last value=1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0

20. Secondary Outcome: Frequency of Participants With Transitions Relative to the Baseline CTC Grade for Neutrophils Based on Last Value on Treatment
Description: Percentage of participants with transitions relative to the baseline CTC grade (version 3) for neutrophils based on last value on treatment.
  Common terminology criteria for adverse events (CTCAE) grade on treatment for neutrophils (CTC version 3). The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE)
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants
  Baseline=0, last value=0 | 100.0 | 66.7 | 100.0 | 66.7 | 91.7 | 66.7 | 100.0 | 100.0 | 100.0 | 83.3 | 69.2 | 100.0
  Baseline=0, last value=1 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 30.8 | 0.0
  Baseline=0, last value=3 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Baseline=1, last value=1 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Baseline=0, last value=2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0
  Baseline=0, last value=4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Baseline=1, last value=0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

21. Secondary Outcome: Frequency of Participants With Transitions Relative to the Baseline CTC Grade for Platelets Based on Worst Value on Treatment
Description: Percentage of participants with transitions relative to the baseline CTC grade (version 3) for platelets based on worst value on treatment.
  Worst Common terminology criteria for adverse events (CTCAE) grade on treatment for platelets (CTC version 3). The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE).
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants
  Baseline=0, worst value=0 | 33.3 | 66.7 | 66.7 | 0.0 | 25.0 | 16.7 | 66.7 | 33.3 | 33.3 | 16.7 | 7.7 | 0.0
  Baseline=0, worst value=1 | 33.3 | 33.3 | 33.3 | 66.7 | 33.3 | 0.0 | 33.3 | 33.3 | 66.7 | 0.0 | 15.4 | 0.0
  Baseline=0, worst value=2 | 0.0 | 0.0 | 0.0 | 33.3 | 8.3 | 66.7 | 0.0 | 0.0 | 0.0 | 33.3 | 15.4 | 33.3
  Baseline=0, worst value=3 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 16.7 | 0.0 | 33.3 | 0.0 | 33.3 | 38.5 | 0.0
  Baseline=1, worst value=1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Baseline=0, worst value=4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 23.1 | 66.7
  Baseline=1, worst value=4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0
  Baseline=1, worst value=0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

22. Secondary Outcome: Frequency of Participants With Transitions Relative to the Baseline CTC Grade for Neutrophils Based on Worst Value on Treatment
Description: Percentage of participants with transitions relative to the baseline CTC grade (version 3) for neutrophils based on worst value on treatment.
  Worst Common terminology criteria for adverse events (CTCAE) grade on treatment for neutrophils (CTC version 3). The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE)
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Percentage of participants
  Baseline=0, worst value=0 | 33.3 | 0.0 | 100.0 | 0.0 | 16.7 | 16.7 | 66.7 | 66.7 | 66.7 | 16.7 | 7.7 | 0.0
  Baseline=0, worst value=1 | 33.3 | 0.0 | 0.0 | 33.3 | 8.3 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 15.4 | 0.0
  Baseline=0, worst value=2 | 33.3 | 33.3 | 0.0 | 0.0 | 25.0 | 0.0 | 0.0 | 0.0 | 33.3 | 16.7 | 15.4 | 0.0
  Baseline=0, worst value=3 | 0.0 | 66.7 | 0.0 | 0.0 | 16.7 | 0.0 | 33.3 | 33.3 | 0.0 | 16.7 | 53.8 | 66.7
  Baseline=0, worst value=4 | 0.0 | 0.0 | 0.0 | 33.3 | 33.3 | 16.7 | 0.0 | 0.0 | 0.0 | 50.0 | 7.7 | 33.3
  Baseline=1, worst value=3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Baseline=1, worst value=4 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

23. Secondary Outcome: Worst CTCAE Grade on Treatment for Platelets
Description: Worst Common terminology criteria for adverse events (CTCAE) grade on treatment for platelets (CTC version 3). The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE).
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Units on a scale
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Units on a scale | 1 (48) | 1 (78) | 1 (94) | 2 (58) | 3 (58) | 3 (95) | 1 (96) | 3 (38) | 1 (65) | 4 (20) | 4 (58) | 4 (53)

24. Secondary Outcome: Worst CTCAE Grade on Treatment for Neutrophils
Description: Worst Common terminology criteria for adverse events (CTCAE) grade on treatment for neutrophils (CTC version 3). The CTCAE scale measures the severity of adverse events which goes from 1 (mild AE) to 5 (death related AE).
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Population: Treated set
Measure: Number; unit: Units on a scale
Arm/Group | V100+Cis60 | V100+Cis75 | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 6 | 3 | 3 | 3 | 6 | 13 | 3
Units on a scale | 2 | 3 | 0 | 4 | 4 | 4 | 3 | 3 | 2 | 4 | 4 | 4

ADVERSE EVENTS:
Time Frame: From first intake of trial drug to last intake of trial drug plus 21 days, up to 441 days
Arm/Group | V200+Cis75 | V300+Cis75 | V300+Cis100 | V350+Cis75 | V100+Car4 | V100+Car5 | V200+Car5 | V300+Car5 | V300+Car6 | V350+Car5 | V100+Cis60 | V100+Cis75
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 6/12 | 3/6 | 1/3 | 0/3 | 1/3 | 1/6 | 6/13 | 2/3 | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 12/12 | 6/6 | 3/3 | 3/3 | 3/3 | 6/6 | 13/13 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V200+Cis75 (N=3) | V300+Cis75 (N=3) | V300+Cis100 (N=12) | V350+Cis75 (N=6) | V100+Car4 (N=3) | V100+Car5 (N=3) | V200+Car5 (N=3) | V300+Car5 (N=6) | V300+Car6 (N=13) | V350+Car5 (N=3) | V100+Cis60 (N=3) | V100+Cis75 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V200+Cis75 (N=3) | V300+Cis75 (N=3) | V300+Cis100 (N=12) | V350+Cis75 (N=6) | V100+Car4 (N=3) | V100+Car5 (N=3) | V200+Car5 (N=3) | V300+Car5 (N=6) | V300+Car6 (N=13) | V350+Car5 (N=3) | V100+Cis60 (N=3) | V100+Cis75 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 8 | 4 | 2 | 3 | 2 | 6 | 12 | 3 | 3 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 9 | 4 | 1 | 1 | 2 | 5 | 11 | 2 | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 7 | 3 | 1 | 1 | 2 | 6 | 8 | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 9 | 4 | 0 | 1 | 1 | 5 | 12 | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 9 | 5 | 1 | 2 | 2 | 5 | 12 | 2 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 4 | 3 | 0 | 0 | 1 | 2 | 6 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Faecal vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 11 | 3 | 0 | 0 | 0 | 3 | 6 | 1 | 2 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 10 | 1 | 0 | 0 | 1 | 2 | 5 | 1 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 8 | 4 | 2 | 1 | 1 | 3 | 8 | 2 | 2 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutrophil count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 7 | 4 | 0 | 1 | 0 | 0 | 6 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Capillaritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.